CLINICAL TRIAL: NCT05104996
Title: The Effect of Discharge Training and Telephone Counseling on Self-Care Agency and Coping And Adaptation Process in Patients Undergoing Coronary Artery Bypass Graft: A Randomized Controlled Study
Brief Title: Discharge Training and Telephone Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Ufuk Kaya, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: EK015/20; Ümran Dal Yılmaz (Other: Near East University)
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Discharge Training and Telephone Counseling for Coronary Artery Bypass Graft Patients
Keywords: coronary artery bypass graft; discharge training; telephone counseling; self-care; coping and adaptation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the first interview, the patients were met and their consent for participation in the study was obtained. Afterwards, The Patient Descriptive Characteristics Form, ESCA and CAPS forms were filled. After this, patients were given discharge training and patient counseling service was provided by telephone for two months after discharge. At the end of two months, the ESCA and CAPS forms were filled again.
  Interventions: Behavioral: Telephone Counseling
- Control Group (No Intervention): In the first interview, the patients were interviewed and their consent was obtained to participate in the study. Then, the Patient Descriptive Characteristics Form, ESCA and CAPS forms were filled. After this, the patients did not undergo any intervention for two months. At the end of two months, the ESCA and CAPS forms were filled again and a copy of the guideline was submitted.

INTERVENTIONS:
Behavioral: Telephone Counseling — The form was used for weekly follow-up of the patients included in the experimental group. Headings were created according to the topics in the training form and/or for other problems and the problems stated by the patients were marked every week. Ongoing or eliminated problems of each patient until the time of next telephone counseling were indicated in the form. General problems in the form included drugs, pain, exercise, wound care, edema, compression socks, corset, nutrition, constipation, bathing, sleep, emergencies, back to work, sexual life, travel, visitors, climbing stairs, alcohol use/smoking, stress/anxiety, check-ups, and other issues.
  Arms: Intervention Group

SUMMARY:
The education and counseling role is one of the independent roles of the nurse. In this context, discharge training and telephone counseling given to patients who underwent coronary artery bypass graft surgery increase the ability of patients to cope with and adapt to their self-care. This study was conducted to determine the effect of discharge training and telephone counseling on self-care agency, coping and adaptation process in patients undergoing coronary artery bypass graft surgery. The study has a randomized controlled, experimental design. Both experimental and control groups consisted of 35 individuals (N=70). Patients in the experimental group were given discharge training and telephone counseling service was given for two months. At the end of the process, data collection forms were administered to both groups for the last time. Necessary ethical approvals were taken and consent was taken from the patients. After the discharge training and telephone counseling given to the experimental group, the mean exercise of self-care agency scale score of the patients increased by 13.94; the mean coping and adaptation processing scale increased by 13.6. The mean exercise of self-care agency scale score of the control group increased by 7.86; the mean coping and adaptation processing score increased by 9.14. The effect size occurred for both groups was statistically significant (p<0.05). Positive results were achieved in the experimental group which received given discharge training and telephone counseling. It is recommended to provide planned discharge training and telephone counseling to patients undergoing coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) is the process of creating a bridge (grafting) to narrowed or clogged coronary arteries using artery and/or vein grafts. Discharge training has many effects such as pain management, reduction of home care visits, reduction of re-admissions to the hospital, acceleration of the recovery process, improvement of self-care agency, reduction of cost, reduction of anxiety level, enhancement of coping and adaptation, and patient satisfaction. Self-care, coping and adaptation remain important in promoting health. Self-care is defined as the decisions and practices made by individuals, who face health concerns, to cope with these concerns, improve their health, and enhance their adaptation. With these improved decisions and practice skills, patients can protect their health more actively. Besides self-care, coping and adaptation are other important issues in patient follow-up. The concept of coping and adaptation is defined as the cognitive and behavioral efforts of the individual to eliminate the necessities and obligations that occur in the inner and outer world, take them under control, and reduce the tension. These efforts may differ according to variables such as family support and spirituality. Patients who are insufficiently informed and not followed up in the postoperative period experience deficits in self-care and difficulties in coping and adaptation. Today, with the increase in the technology use, patient counseling by telephone can be provided for patient follow-up at home, monitoring drug side effects, counseling, sudden situations, appointment reminder, evaluation of the effectiveness of discharge training, determining training needs, performance evaluation, providing communication between hospital and home, increasing participation in training, improving self-care, increasing quality of life, ensuring coping and adaptation. Postoperative care outcomes and the patient's medical condition can be improved by ensuring continuity in telephone counseling. Postoperative mobile health applications are important in terms of evaluating changes, that may occur in the home environment, on time. Today, the rapid development of medicine and technology and the development of products that facilitate monitoring patients can help individuals who have undergone CABG surgery through telephone counseling and patient training. Training and telephone counseling services may reduce the number of hospital admissions, increase self-care agency, improve the quality of life, and enhance coping and adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone CABG surgery,
* Being able to speak, read and write in Turkish,
* Not having a visual, hearing, physical, and mentally disability,
* Being aged over 18.

Exclusion Criteria:

* Being unable to speak, read and write in Turkish,
* Having a visual, hearing, physical, and mentally disability,
* Being aged under 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Exercise of Self-Care Agency Scale (ESCA) | 2 months
  The scale was developed by Kearney and Fleicher in 1979 and is originally a 43-item English form. The five-point Likert-type questionnaire aims to determine the ability of individuals to care for themselves and their self-care agency. The scale consists of statements scored from 0 to 4. It consists of a scale of 'very uncharacteristic of me' (0), 'somewhat uncharacteristic of me' (1), 'uncertain' (2), 'somewhat characteristic of me' (3), and 'very characteristic of me' (4) in each statement. Eight negative statements on the scale (3, 6, 9, 13, 19, 22, 26, and 31) are scored reversely. The lowest score obtainable from the scale is 35 and the highest score is 140.
Coping and Adaptation Processing Scale (CAPS) | 2 months
  It is theoretically based on the Roy Adaptation Model and concepts related to its cognitive process. The scale consists of subscales such as troubleshooting and focusing, physical and conclusion, attention process, systematizing process, learning and establishing relationship. The number of items in the subdimensions is as follows: 'troubleshooting and focusing' involves 10 items; 'physical and conclusion' involves 14 items: 'attention process' involves 9 items; 'systematizing process' involves 6 items; 'learning and establishing relationship' involves 8 items. Items are scored on a Likert-type scale: 'never', 'rarely', 'sometimes', and 'always'.

SECONDARY OUTCOMES:
Telephone Counseling Patient Follow-up Form | 2 months
  The form was used for weekly follow-up of the patients included in the experimental group. Headings were created according to the topics in the training form and/or for other problems and the problems stated by the patients were marked every week. Ongoing or eliminated problems of each patient until the time of next telephone counseling were indicated in the form. General problems in the form included drugs, pain, exercise, wound care, edema, compression socks, corset, nutrition, constipation, bathing, sleep, emergencies, back to work, sexual life, travel, visitors, climbing stairs, alcohol use/smoking, stress/anxiety, check-ups, and other issues.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Naveed A, Azam H, Murtaza HG, Ahmad RA, Baig MAR. Incidence and risk factors of Pulmonary Complications after Cardiopulmonary bypass. Pak J Med Sci. 2017 Jul-Aug;33(4):993-996. doi: 10.12669/pjms.334.12846. PMID 29067080
- [Result] Yuroong A, Asdornwised U, Pinyopasakul W, Wongkornrat W, Chansatitporn N. The Effectiveness of the Transitional Care Program Among People Awaiting Coronary Artery Bypass Graft Surgery: A Randomized Control Trial. J Nurs Scholarsh. 2021 Sep;53(5):585-594. doi: 10.1111/jnu.12673. Epub 2021 May 19. PMID 34013579
- [Result] Williams B. Supporting self-care of patients following general abdominal surgery. J Clin Nurs. 2008 Mar;17(5):584-92. doi: 10.1111/j.1365-2702.2006.01857.x. PMID 18279291
- [Result] Jerant AF, Azari R, Martinez C, Nesbitt TS. A randomized trial of telenursing to reduce hospitalization for heart failure: patient-centered outcomes and nursing indicators. Home Health Care Serv Q. 2003;22(1):1-20. doi: 10.1300/J027v22n01_01. PMID 12749524
- [Derived] Kaya U, Dal Yilmaz U. Ideal Suggestions for Discharge Training and Telephone Counseling of Patients With Coronary Artery Bypass Graft Surgery: A Randomized Controlled and Experimental Study. J Korean Med Sci. 2022 Sep 5;37(35):e269. doi: 10.3346/jkms.2022.37.e269. PMID 36065653